CLINICAL TRIAL: NCT02084251
Title: Safety, Tolerability and Pharmacokinetics of Single Dose of PB-119 in Healthy Volunteers
Brief Title: Clinical Trial for PB-119 in Healthy Subjects (Phase I)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PegBio Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: ICP-I-2013-08
Record Dates: First submitted 2014-03-09; First posted 2014-03-11 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Type II Diabetes
Keywords: safety,; pharmacokinetics,; Long acting GLP-1 analogue
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Exenatide analogue, Injection (Experimental): PB-119 will be administered once weekly subcutaneously at dosage of 2μg、5μg、10μg、25μg、50μg、100μg、200μg or 400μg.
  Interventions: Drug: PB-119

INTERVENTIONS:
Drug: PB-119

SUMMARY:
GLP-1 analogues have been widely used because of their unique advantages (no risk of hypoglycemia) due to their glucose dependent mechanism. Due to the short half-life of peptide in plasma, peptides have to be administered frequently (i.e. BID for Byetta, with Exenatide as API).To improve the patients compliance and reduce potential adverse events associated with GLP-1 analogues, a long acting GLP-1 analogue (PB-119), which may be administered once weekly, was developed by PegBio Inc. In order to provide rational for dosage range to be studied in Phase Ib, the safety profile, tolerance, and pharmacokinetic behavior of PB-119 in healthy subjects will be studied in this randomized, controlled dose escalating trial.

ELIGIBILITY:
Inclusion Criteria:

* Male or female volunteers, ages: between 18-45;
* Body weight： female >= 45kg, male >=50kg, BMI >=19-24kg/m2
* Physical examination, blood routine, urine routine, liver and kidney function and related laboratory tests are normal or slightly abnormal but not clinically significant;
* Read, agree, and sign the informed consent;
* Be able to communicate with the investigator and finish the study according to the protocol.

Exclusion Criteria （anyone or more of the following):

* Allergic to the API or excipients used (citric acid, mannitol, Meta-Cresol);
* Experiencing clinically significant disease or surgery within 4 weeks before the study;
* Clinically significant disease history in systems including cardiovascular system, endocrine system, neutral system, immunology system, psychiatry，metabolic disorder;
* Disease history of gastrointestinal tract, liver, and kidney (for example, the Partial resection surgery in GI tract, liver, or kidney);
* Fever history within 3 days of the screening;
* Clinical significant abnormality found in laboratory tests (blood, urine routine test) within 2 weeks before study;
* ECG or vital signs is clinically significant abnormality as judged by the Investigator( systolic blood pressure <90mmHg or ≥140mmHg; diastolic blood pressure<60mmHg or ≥90mmHg; heart rate <50bpm or >100bpm);
* Antibody test for HIV, BsAg, C hepatitis, or Microspironema pallidum positive;
* Alcoholics or drink frequently within 6 months of trial (more than 14 unit of alcohol, in which 1 unit is 360mL beers, or 45 ml wine with 40% alcohol content, or 150mL port wine;
* Addicted to cigarette, tea, coffee or drugs;
* Have specific requirement for diets (or allergic to any food);
* Have been administered in the past 2 weeks with any drug (such as antibiotics, anticoagulant, diuretics) that might interfere the PK profile of drug/drug candidate to be used in this study;
* Participated in any clinical trial in the past 3 months;
* Donated blood of more than 360 ml in the past 3 months;
* Plan to be pregnant herself or his spouse in the next 6 months;
* Females administered with any oral contraceptive 30 days before the study or during the study;
* Females dosed with long acting estrogen or progestin (injections or implant) 6 months before the study or during the study;
* Females at childbearing age that had unprotected intercourse 14 days before the study or will have during the study;
* Female who is pregnant or nursing;
* Anybody who might not be able to complete the study, or considered not appropriate by the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2014-02; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Safety/Adverse Event Outcome Measure | Up to 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Lv, Doctor, Principal Investigator — No.1 Hospital of Peking University
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Cui H, Zhao CY, Lv Y, Wei MJ, Zhu Y, Li Y, Xia YH, Liu Y, Tian JH, Zhang P. Safety, Tolerability and Pharmacokinetics of Single Dose Polyethylene Glycolated Exenatide Injection (PB-119) in Healthy Volunteers. Eur J Drug Metab Pharmacokinet. 2020 Jun;45(3):361-369. doi: 10.1007/s13318-020-00605-9. PMID 32006325